CLINICAL TRIAL: NCT04476199
Title: Phase II Study on Venetoclax (VEN) Plus Decitabine (DEC) (VEN-DEC) for Elderly (≥60 <75years) Patients with Newly Diagnosed Acute Myeloid Leukemia (AML) Elegible for Allogeneic Stem Cell Transplantation (allo-SCT)
Brief Title: Venetoclax and Decitabine Assessment in Patients (≥60 - <75 Years) with Newly Diagnosed AML Eligible for Allo-SCT
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Italiano Trapianto di Midollo Osseo (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GITMO-VEN-DEC
Record Dates: First submitted 2020-07-02; First posted 2020-07-20 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia; Allogenic Stem Cell Transplant
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — venetoclax; Decitabine

STUDY DESIGN:
Intervention Model Description: These patients may undergo allo-SCT after 2 - 4 cycles of VEN-DEC
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment with VEN-DEC (Experimental): Venetoclax will be given with a 3-day ramp up beginning with 100 mg dose on Day 1, with 200mg on Day 2, to reach the final dose of 400 mg on Day 3 of Cycle 1. Venetoclax will be continued at 400 mg daily. Tumor lysis prophylaxis will be administered from day -4, cycle 1 (oral uric acid reducing agent and hydration with at least 1.5 L/day).Decitabine will be administered at the dose of 20 mg/sqm intravenously from day 1 to day 5 every 28 days (VEN-DEC) for 2 cycles.
  Interventions: Combination Product: Venetoclax and Decitabine

INTERVENTIONS:
Combination Product: Venetoclax and Decitabine — The prognosis of acute myeloid leukemia (AML) patients aged over 60 years is poor and allogeneic stem cell transplantation (allo-SCT) is the only curative option.The association VEN-DEC is a promising combination therapy for AML elderly patients who are fit and eligible for allo-SCT.

SUMMARY:
This trial is a no profit, prospective, phase II, multicentre, non-randomised, uncontrolled, single group assignment, open label study to evaluate the safety and efficacy of the "chemo-free" combination Venetoclax plus Decitabine (VEN-DEC) as "bridge" to allo-SCT in elderly (≥ 60 - < 75 years) AML patients. The primary objective is to evaluate the proportion of elderly (≥60 - <75 years) patients with newly diagnosed AML, eligible for allo-SCT, treated with the "chemo-free" combination Venetoclax plus Decitabine (VEN-DEC) who get allo-SCT in CR/Cri/MLFS.

DETAILED DESCRIPTION:
This trial is a no profit, prospective, phase II, multicentre, non-randomised, uncontrolled, single group assignment, open label study to evaluate the proportion of elderly (≥60 - <75 years) patients with newly diagnosed AML, eligible for allo-SCT, treated with the "chemo-free" combination Venetoclax plus Decitabine (VEN-DEC) who get allo-SCT in CR/CRi/MLFS, organized under the auspices of the Gruppo Italiano TRapianti di Midollo Osseo (GITMO) that involves the prinicipla centres active in transplantation of any kind of stem cells in Italy. The target for this study is 100 patients.

Biologic characterization of AML will be performed at each participating Center by flow cytometry, cytogenetics and RT-qPCR on target genes (FLT3, NPM1A, WT1,) at disease onset. MRD monitoring will be performed at each participating Center by flow cytometry, cytogenetics and RT-qPCR (routine assessment) at the time of CR/CRi/MLFS before allo-SCT and during follow up (at least 4 timepoints: +100 days, +180 days, +1 year and +2 years from allo-SCT).

Genomic analysis by NGS gene-panel (Sophia Genetics) exploring the mutational status of the genes involved in of AML will be centralized in Brescia Laboratory at the enrollment into the study (diagnosis) and at the time of no response (PR/NR), before allo-SCT in patients in CR/CRi/MLFS and in case of relapse, at any time.

Primary Objectives To evaluate the proportion of elderly (≥60 - <75 years) patients with newly diagnosed AML eligible for allo-SCT treated with the "chemo-free" combination Venetoclax plus Decitabine (VEN-DEC) who get allo-SCT in CR/CRi/MLFS.

Secondary Objectives

* Incidence and severity of adverse drug reactions (ADR) classified by System Organ Class (SOC) and preferred term (PT) from start treatment with Ventoclax and Decitabine to allo-SCT
* Efficacy of VEN-DEC combination
* Evaluation of the outcome of allo-SCT in term of:1) Incidence of graft failure at day +30, +100 from allo-SCT2) Incidence of Non-Relapse Mortality (NRM) at day +100, 1 year and 2 years from allo-SCT3) Incidence and severity of acute GVHD at day +100 from allo-SCT4) Incidence and severity of chronic GVHD at 1 year and 2 years from allo-SCT5) Probability of GRFS (GVHD free, relapse free survival) at 1 and 2 years from allo-SCT
* Relapse incidence (RI) at 1 year and 2 years from allo-SCT
* Disease-free survival (DFS) at 1 and 2 years from allo-SCT
* Overall Survival (OS) at 1 and 2 years from allo-SCT
* Correlation of immunophenothype, cytogenetic, molecular and NGS-genomic profiles with sensitivity (CR - CRi - MLFS) or resistance (PR/NR) to "chemo-free" combination Venetoclax plus Decitabine (VEN-DEC)
* Correlation of immunophenothype, cytogenetic, molecular and NGS-genomic profiles with the outcome of allo-SCT in terms of NRM, probability of RI, DFS, OS.

This study has 2 endpoints

Primary Endpoint Proportion of elderly (≥60 - <75 years) patients with newly diagnosed AML eligible for allo-SCT treated with the "chemo-free" combination Venetoclax plus Decitabine (VEN-DEC) who get allo-SCT in CR/CRi/MLFS.

Secondary Endpoints

* Efficacy of VEN-DEC combination
* Cumulative incidence of graft failure at +30 days, +100 days from transplant
* Outcome of allo-SCT in term of NRM at day +100, 1 year and 2 years from allo-SCT
* Cumulative incidence and severity of acute GvHD at 100 days after transplant
* Cumulative incidence and severity of chronic GvHD at 1 and 2 years post transplant
* RI at 1 and 2 year after transplantation from days of transplant.
* OS at 1 and 2 years post transplant
* DFS at 1 and 2 years post transplant
* 1 and 2 year probability of GRFS
* Correlation of immunophenothype, cytogenetic, molecular and NGS-genomic profiles with sensitivity (CR - CRi - MLFS) or resistance (PR-NR) to "chemo-free" combination Venetoclax plus Decitabine (VEN-DEC)
* Correlation of immunophenothype, cytogenetic, molecular and NGS-genomic profiles with the outcomes of allo-SCT: NRM, RI, DFS, OS.

Biologic characterization of AML will be performed at each participating Center by flow cytometry, cytogenetics and RT-qPCR on target genes (FLT3, NPM1A, WT1,…) at disease onset. MRD monitoring will be performed at each participating Center by flow cytometry, cytogenetics and RT-qPCR (routine assessment) at the time of CR/CRi/MLFS, before allo-SCT and during follow up (at least 4 timepoints: +100 days, +180 days, +1 year and +2 years from allo-SCT).Genomic analysis by NGS gene-panel (Sophia Genetics) exploring the mutational status of the genes involved in of AML will be centralized in Brescia Laboratory at the enrollment into the study (diagnosis) and at the time of no response (PR/NR), before allo-SCT in patients in CR/CRi/MLFS and in case of relapse, at any time.

Venetoclax will be given with a 3-day ramp up beginning with 100 mg dose on Day 1 to reach the final dose of 400 mg on Day 3 of Cycle 1. Venetoclax will be continued at 400 mg daily. Tumor lysis prophylaxis will be administered from day -4, cycle 1 (oral uric acid reducing agent and hydration with at least 1.5 L/day).

Decitabine will be administered at the dose of 20 mg/sqm intravenously from day 1 to day 5 every 28 days (VEN-DEC) for 2 cycles. The response will be assessed after the 2nd Cycle VEN-DEC according to ELN criteria. In case of CR/CRi/MLFS, patients will undergo allo-SCT within 2 months. A maximum of two additional VEN-DEC cycles is permitted while waiting for allo-SCT. In case of NR or PR after the 2nd Cycle VEN-DEC, two additional cycles of VEN-DEC will be administered and patients achieving CR/CRi/MLFS will undergo allo-SCT as soon as possible (within 2 months). Patients with NR or PR will be treated according to single center policy, including also allo-SCT.

Patients achieving Morphologic Leukemia-free State (MLFS) will be considered responsive patients, since the percentage of BM blast cells is < 5%. These patients may undergo allo-SCT after 2 - 4 cycles of VEN-DEC.Granulocyte colony stimulating factor (G-CSF) will be allowed during VEN-DEC in case of febrile neutropenia. Whenever clinically indicated, G-CSF use has to be notified tin the CRF.

Population for analysis The population for analysis in this trial will be the Intent to Treat (ITT) population. All patients who have received at least one therapeutic dose of study medications will be included in the ITT analysis.

Sample size calculation The study is designed as a Simon optimal two-Stage Phase II clinical trial, including a planned futility check: after enrollment of the first 30 patients the Investigator will pause for the futility check is at that time point the target 4 patients will not yet be admitted to allo-SCT. Based on the current literature, less than 10% of elderly (>60 <75 years) AML patients can be submitted to allo-SCT, due to no-response to induction conventional chemotherapy (NR or PR) and /or to treatment toxicity. Therefore, to test the null hypothesis (conventional chemotherapy) that p ≤0.10 versus the alternative (VEN-DEC) that p ≥0.20, the expected sample size is 89 patients, with a probability of early termination of 0.647, when true proportion is 0.1. Alpha error is 0.0478 and beta value 0.1982. If there are 3 or fewer patients submitted to allo-SCT in the first 30 enrolled patients, the trial will be terminated for futility. Otherwise, considering an overall 12% of drop-out rate, 70 additional patients will be accrued for a total of 100 patients: in the second stage 70 patients will only be enrolled if at least 4 patients of the first stage undergo allo-SCT. The null hypothesis will be rejected if 14 of more patients treated with VEN-DEC will be submitted to allo-SCT in CR/CRi/MLFS.

The study is considered completed when the 100th patient will be enrolled. It is planned to complete the total enrollment (100 patients) in 18 months, starting from the first patient enrolled.

The follow-up according to the protocol is 2 years for each patient from the day of enrollment. In the transplanted patients the pre-transplant period will be followed by 2 years post-transplant follow-up

The study will be performed in 4 years from the first patient enrolled according to the following times:

18 moths for enrollment (from the first patient) and for database completion and cleaning 24 months of follow up. In the transplanted patients the pre-transplant period will be followed by 2 years post-transplant follow-up 6 months for statistical analysis, drafting of the final report and paper.

The study will be conducted in accordance with the ethical principles derived from the Declaration of Helsinki, the CGP and regulations.

Before starting the study, the protocol will be sent to the Ethics Committee, in accordance with the current legislation on interventional study.

The protocol has been written and the study will be conducted according to the International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use Harmonized tripartite Guideline for GCP, issued by European Union. IRB approval must be obtained prior to the starting of the trial. ICF must be submitted to appropriate authority or IRB together with clinical protocol for written approval.

ELIGIBILITY:
Inclusion Criteria:

* • Patients >60 <75 years of age

  * Diagnosis of AML eligible for allo-SCT from any donor
  * High- and Intermediate-Risk ELN
  * WBC <25x109/L (Hydroxyurea is permitted to meet this criterion)
  * adequate hepatic function (bilirubin ≤2 UNL; ALT/AST ≤2,5 UNL)
  * adequate renal function (creatinine clearance ≥50 ml/min)
  * ECOG Performance Status < 2
  * Males enrolled in the study with partners who are women of childbearing potential, must be willing to use an acceptable barrier contraceptive method during the trial.
  * Women of childbearing potential must use highly effective contraception for at least 1 month after the last dose of VEN and for however long the EU SmPC says for DEC
  * Willing and able to comply with all of the requirements and visits in the protocol.
  * Written and signed informed consent.

Exclusion Criteria:

* • Previous treatment for AML (Hydroxyurea is allowed) or for an antecedent Myelodysplastic Syndrome (MDS).

  * Absence of informed consent
  * AML patients with t(15;17); t(8;21); inv(16)
  * Subject has known active CNS involvement with AML.
  * Low Risk ELN
  * grade >2 NCI-CTCAE (v. 5) adverse events at the time of enrollment
  * Serious organ dysfunction: left ventricular ejection fraction < 40%, FEV1, FVC, DLCO (diffusion capacity) <40% of predicted, LFT > 5 times the upper limit of normal, or creatinine clearance < 40 ml/min.
  * The evidence of HBV or HCV active infection (HBV DNA HCV RNA positive test).
  * Patients with HIV infection
  * Current uncontrolled infections
  * Patients with other life-threatening concurrent disease
  * Subjects with known hypersensitivity to any of the component medication
  * Subject has a history of other malignancies within 2 years prior to study entry, with the exception of:
* Adequately treated in situ carcinoma of the cervix uteri or carcinoma in situ of breast;
* Basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin;
* Previous malignancy confined and surgically resected (or treated with other modalities) with curative intent. • Participation in another clinical trial within 1 month before the start of this trial

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2023-02-03 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Response to VEN-DEC chemo-free combination (ELN Guidelines) | At the end of cycle 2 (each cycle is 28 days)
  response to VEN-DEC induction will be assessed on bone marrow according to the ELN Guidelines (13), as following: - CR without minimal residual disease (CR-MRD neg); (Complete Remission ) bone marrow blasts 5%) - CR remission with incomplete hematologic recovery (CRi): Morphologic Leukemia-free State (MLFS) Partial Remission (PR): All hematologic criteria of CR; decrease of bone marrow blast percentage to 5% to 25%; and decrease of pretreatment bone marrow blast percentage by at least 50%; - Primary refractory disease/Non response (NR): No CR or CRi after 2 courses of VEN-DEC; excluding patients with death in aplasia or death due to indeterminate cause;
Allo-SCT | 18 months from 1st enrolled patient
  Proportion of patients who undergo to allo-SCT in first CR/CRi/MLFS
Allo-SCT Engraftment | up to 24 weeks
  Percentage of patients with Neutrophil engraftment and percentage of patients with platelet engraftment
Overall Survival (OS) | at 2 year post transplant
  at 2 year post transplant. OS is defined as the time from transplant to the date of death due to any cause or to the last date the patient was known to be alive (censored observation) or to the date of the data cut-off for final analysis
Cumulative incidence of Non-Relapse Mortality | at 100 days
  NRM is defined as death due to any other cause than progression of malignancy after allogeneic stem cell transplantation. Cumulative incidence will be estimated at 100 days
Cumulative incidence of Non-Relapse Mortality | at 180 days
  NRM is defined as death due to any other cause than progression of malignancy after allogeneic stem cell transplantation. Cumulative incidence will be estimated at 180 days
Cumulative incidence of Non-Relapse Mortality | at 365 days
  NRM is defined as death due to any other cause than progression of malignancy after allogeneic stem cell transplantation. Cumulative incidence will be estimated at 365 days

CONTACTS AND LOCATIONS:
Overall Officials: Domenico Russo, MD, Principal Investigator — Spedali Civili Brescia
Locations (25):
- Italy (25):
  - USD, Trapianti di Midollo osseo, Azienda Spedali Civili di Brescia, Brescia, Brescia
  - Unità Terapia Intensiva Ematologica e terapia cellulari - casa della sofferenza, San Giovanni Rotondo, Foggia
  - UO Ematologia e TMO - Ospedale C. Panico, Tricase, Lecce
  - Ospedale San Gerardo, Monza, Monza
  - Clinica di Ematologia. AOU Ospedali Riuniti di Ancona, Ancona
  - UOC di Ematologia, Ospedale C e G Mazzoni, Ascoli Piceno
  - U.O. Ematologia con Trapianto, Policlinico di Bari, Bari
  - Ospedale Seragnoli Malpighi, Bologna
  - Ospedale Policlinico di Catania, TMO, Catania
  - Struttura Complessa di Ematologia, Azienda Ospedaliera Santa Croce e Carle, Cuneo
  - Terapie Cellulari e Medicina Trasfusionale, Ospedale Careggi, Florence
  - UO Ematologia, Programma Trapianti IRCCS Ospedale Policlinico San Martino, Genova, Genova
  - Centro Trapianto Fondazione IRCCS Cà Granda - Osp. Maggiore, Milan
  - Div. di Ematologia e TMO, Istituto Nazionale Tumori, Milan
  - Div. di Ematologia, Talamona, Osp. Niguarda, Ca-Granda, Milan
  - Istituto Clinico Humanitas, Oncologia ed Ematologia, Milan
  - Unità Operativa di Ematologia e Trapianto Midollo Osseo (UTMO), Ospedale San Raffaele di Milano, Milan
  - UOSC Ematologia con Trapianto CSE, AORN A. Cardarelli, AORN Cardarelli, Napoli
  - CTMO Osp. V. Cervello Azienda Ospedaliera Ospedali Riuniti Villa Sofia Cervello, Palermo
  - Dip.di Ematologia, Osp. Civile di Pescara, Unità di Terapia Intensiva Ematologica per il Trapianto Emopoietico, Pescara
  - CTMO Centro Unico, Regionale Trapianti di Cellule Staminali e Terapie Cellulari, "A. Neri", Grande Osp. Bianchi, Melacrino Morelli, Reggio Calabria
  - Policlinico Tor Vergata, Roma
  - A.O.U. Citta della Salute e della Scienza, Torino
  - UOC di Ematologia, Osp. dell'Angelo, Venezia
  - Div. di Ematologia - Unità di TMO e Oncoematologia Pediatrica Policlinico GB Rossi, Verona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Russo D, Polverelli N, Bernardi S, Santarone S, Farina M, Borlenghi E, Onida F, Castagna L, Bramanti S, Carella AM, Sorasio R, Martino M, Alati C, Olivieri A, Beltrami G, Curti A, Vetro C, Leotta S, Mancini V, Terruzzi E, Bernardi M, Galieni P, Musto P, Cerretti R, Giaccone L, Skert C, Radici V, Vezzoli M, Calza S, Leoni A, Garuffo L, Bonvicini C, Pellizzeri S, Malagola M, Ciceri F. Venetoclax plus decitabine as a bridge to allogeneic haematopoietic stem-cell transplantation in older patients with acute myeloid leukaemia (VEN-DEC GITMO): final report of a multicentre, single-arm, phase 2 trial. Lancet Haematol. 2024 Nov;11(11):e830-e838. doi: 10.1016/S2352-3026(24)00241-2. Epub 2024 Sep 20. PMID 39312920